CLINICAL TRIAL: NCT05313191
Title: Prospective Evaluation of Pencil Beam Scanning Proton Therapy for Previously Irradiated Tumors
Acronym: ReRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The New York Proton Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYPC ERC# 2019-002
Record Dates: First submitted 2022-03-21; First posted 2022-04-06 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: CNS Cancer; Head and Neck Cancer; GI Cancer; Gynecologic Cancer; Prostate Cancer; Thoracic Cancer; Breast Cancer
Keywords: Reirradiation; Cancer; Proton Therapy; Radiation Therapy
MeSH Terms: conditions — Central Nervous System Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase: Registry, Phase I, Phase II Study Design/Methodology: Cohort-defined, single arm prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (8):
- Cohort 1: Central Nervous System (Experimental): Group 1 Definitive Reirradiation Phase II
  * Patients w/history of intracranial or spinal (extradural, intradural, and/or intramedullary) CNS tumors for which radiation therapy was prev. delivered either to gross disease or in the postoperative setting
  * Min. 6 month interval b/w RT courses
  * Overlap of prior RT field (50% IDL)
  * Subgroup analysis: receipt of surgery for recurrence/second IC tumor; concurrent ST; tumor histology
  Group 2 CNS Reirradiation Registry
  * Patients for whom a repeat course of RT to the CNS is indicated for recurrent disease or secondary primary
  * Postop or intact setting
  * Min. 6 month interval b/w RT courses
  * Overlap of prior RT field (50% IDL)
  * Histologically/clinically documented recurrent CNS tumor (benign or malignant)
  * Glioblastoma (histologic or molecular including IDH wildtype)
  * Astrocytoma (molecular IDH1 mutant)
  * Oligodendroglioma (molecular 1p19q co deleted)
  * Meningioma
  * Ependymoma
  * Chordoma/chondrosarcoma
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 2: Head/Neck (Experimental): Group 1 Full Dose Reirradiation Phase II
  * Patients w/history of HNC for which RT was delivered definitively, now with recurrence to h/n amenable to full dose reRT
  * Gross unresected disease or PORT 2/2 RF
  * Received at least 40 Gy overlapping w/new target region
  * Min. 6 month interval b/w RT courses
  * Overlap of prior RT field (50% IDL)
  * Subgroup analysis: surgery, HPV status, concurrent ST
  Group 2 Early (<6months for prior RT) Palliative H/N ReRT Phase I
  * Patients w/history of HNC for which RT was delivered definitively/adjuvant setting, now with biopsy proven recurrence to h/n with indication for palliative RT
  * At least 30 Gy prior RT overlapping with new treatment volume
  * <6 month interval between RT courses
  Group 3 Head/Neck ReRT Registry
  * Patients w/history of HNC for which RT was delivered now with recurrence/secondary primary requiring reRT
  * Postop or definitive
  * Prior RT dose at least 30 Gy overlapping w/new treatment volume
  * Min.6 month interval b/w RT courses
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 3: Breast (Experimental): Group 1 Partial Breast Reirradiation (Phase II)
  * Patients with a history of breast cancer s/p BCT, now with small (≤3cm), unicentric, ipsilateral breast cancer recurrence receiving repeat BCT
  * Node negative
  * Negative margins
  * No LVI
  * Lumpectomy cavity:whole breast <30%
  * Minimum 1 year interval between RT courses
  Group 2: Regional LN and Breast/CW ReRT (Phase II)
  * Patients with a history of breast cancer s/p RT , now with recurrence or new primary with indication for reirradiation to the breast/chest wall and regional LN
  * Minimum 1 year interval between RT courses
  * Negative metastatic workup (PET/CT or CT C/A/P + bone scan)
  * Excludes concurrent chemotherapy
  Group 3: Breast Reirradiation Registry
  * Patients with a history of breast cancer s/p RT , now with recurrence or new primary breast cancer with indication for reirradiation
  * Some overlaps of dose with prior RT course
  * Negative metastatic workup (PET/CT or CT C/A/P + bone scan)
  * Excludes concurrent chemotherapy
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 4: Thoracic (Experimental): Group 1: Definitive Reirradiation for Locally Advanced Disease
  * Single arm, prospective, phase II study
  * Patients with a history of lung cancer s/p definitive RT , now with local recurrence of new primary centrally located and w/I 50% IDL of prior RT field
  * Definitive reRT concurrent systemic therapy
  * Adequate pulmonary function defined as an FEV1 of >35% (with or without bronchodilator) within 90 days prior to registration
  * Minimum 6 month interval between RT courses
  * Negative metastatic workup
  Group 2: Thoracic Registry Study
  * Registry design
  * Patients with histologically confirmed thoracic malignancy (NSCLC, SCLC , mesothelioma, thymoma, carcinoid, intrathoracic sarcoma) with prior thoracic RT
  * Minimum 3 month interval between RT courses
  * Negative metastatic workup
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 5: Gastrointestinal (Experimental): Group 1 Esophagus & GEJ Reirradiation Phase II
  * Patients w/history of E/GEJ cancer s/p RT, now w/recurrent/new primary nonmetastatic E/GEJ cancer for which salvage RT is recommended
  * Negative metastatic workup
  Group 2 Liver Reirradiation Phase II
  * Patients w/history of HCC, cholangiocarcinoma or liver mets (any histology), s/p prior EBRT, now with in field recurrence/new primary/met, for which definitive reRT is recommended
  * CTP A or B7
  * Excl. prev. Y 90/radioembolization
  * Allow prior TACE
  * Overlap w/50% IDL prior RT
  * Adequate bone marrow function
  Group 3 Lower GI Reirradiation Phase II
  * Patients w/history of rectal/anal cancer s/p RT now w/recurrent/new primary nonmetastatic rectal/anal cancer for whom salvage RT is recommended +/ chemotherapy
  * Negative metastatic workup (PET/CT or CT C/A/P)
  Group 4 GI Reirradiation Registry
  •Patients w/histologically document recurrent or new GI malignancy with prior history of RT w/overlap of current RT volume by the 50% IDL
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 6: Genitourinary (Experimental): Group 1 Locally recurrent prostate cancer w/in prev. radiation field Phase II
  * Patients w/recurrent prostate adenocarcinoma w/in prev. irradiated field w/indication for repeat course of radiation
  * Min. 1 year interval b/w RT courses
  * Prostate gland or recurrent tumor <100 cc or 6 cm in largest dimension
  * No persistent grade 2+ toxicity from prior radiation
  * Negative metastatic workup (bone scan, CT scan or PSMA/axumin scan
  Group 2 Regional prostate cancer recurrence adjacent to the previous field Phase II
  * Patients w/recurrent prostate adenocarcinoma beyond prior RT field (outside 50% IDL) but w/in pelvis)
  * Min.1 year interval b/w RT courses (EBRT or brachy)
  * No persistent grade 2+ toxicity from prior radiation
  Group 3 Prostate Reirradiation Registry
  * Patients w/recurrent prostate adenocarcinoma (prostate gland, postop bed, or pelvi c LN) who require RT to the prostate or pelvis in the setting of prior pelvis RT
  * No DM
  * Concurrent chemotherapy excl.
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 7: Gynecological (Experimental): Group 1: Locally recurrent gynecological cancer within previous field
  * Single arm, prospective, phase II study design
  * Patients with history of gyn cancer for which definitive or adjuvant/salvage PORT was given, now with recurrence within 50% IDL recommended for radiotherapy
  * At least 1 year between RT courses
  * No persistent grade 3+ toxicity from prior RT
  * Concurrent chemotherapy excluded
  * Uncontrolled or widely metastatic disease
  * Life expectancy >6 months
  Interventions: Radiation: Pencil Beam Scanning Proton Therapy
- Cohort 8: Registry (No Intervention): * Registry design
  * Any cancer patient for whom RT is indicated in the setting of prior RT and do not meet eligibility criteria for other cohorts
  * Overlap of 50% IDL of current treatment volume with prior RT field

INTERVENTIONS:
Radiation: Pencil Beam Scanning Proton Therapy — Use of Pencil Beam Scanning Proton Therapy compared with historical outcomes using photon therapy for the reirradiation of recurrent or new primary malignancies
  Arms: Cohort 1: Central Nervous System; Cohort 2: Head/Neck; Cohort 3: Breast; Cohort 4: Thoracic; Cohort 5: Gastrointestinal; Cohort 6: Genitourinary; Cohort 7: Gynecological

SUMMARY:
The goal of this clinical research trial is to study the use of differing investigational doses and scheduling for Proton Therapy for tumors previously treated with radiation therapy. Generally, when patients are first treated for cancer with radiation therapy, they are treated with traditional photon (or x-ray) radiation therapy, which uses high-energy waves to kill tumor cells. In some cases, the cancer either returns or a new tumor can present in a different part of the body. With the usual radiation treatment, the photon beams travel all the way through the body. As a result, healthy tissues in front of and behind the tumor are exposed to radiation. Physicians who treat these cases where the tumor has returned often use a much lower dose of radiation to prevent patients from experiencing serious and long-term side-effects. This dose is often not strong enough to destroy the cancerous tumor. Alternatively, they may also treat a smaller area than would be indicated for complete tumor eradication, again in an attempt to prevent serious and long-term toxicities, but at the cost of optimally treating the cancer. Proton therapy, however, may offer a chance to safely deliver a more effective dose and volume of radiation as it is more targeted and can spare healthy tissues surrounding the tumor.

The reason we are conducting this research study is to look at whether Proton therapy can be a better way to treat reoccurring tumors in patients who have previously received radiation therapy to the same area, compared to treatment approaches used to date.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Patient provides study specific informed consent prior to study entry.
* Documented history and physical exam within 90 days prior to registration.
* ECOG PS 0, 1, or 2 within 90 days prior to registration

Exclusion Criteria:

* Non malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow up.
* Prior invasive non study malignancy unless disease free for ≥ 3 years

  * Non melanoma skin cancer, low risk prostate cancer, well differentiated thyroid cancers, in situ carcinomas of the oral cavity, cervix, and other organs, and tumors that are not thought to impact the life expectancy of the patient are permissible.
* History of active connective tissue disorder (i.e., systemic lupus erythematosus, scleroderma), dermatomyositis, xeroderma pigmentosum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To determine the cumulative rate of CTCAE v5.0 Grade ≥3 acute and late treatment related adverse events within 1 year of definitive reirradiation completion using proton therapy for recurrent or second primary tumor. | 5 years

SECONDARY OUTCOMES:
To determine the 1 year freedom from local failure. | 1 year
To determine the 1 year freedom from progression free survival. | 1 year
To determine the 1 year freedom from overall survival. | 1 year
To determine the acute cumulative rate of CTCAE v5.0 Grade ≥3 treatment related adverse events at 90 days of reirradiation completion. | 90 days
To determine the late cumulative rate of CTCAE v5.0 Grade ≥3 treatment related adverse events at 2 years of reirradiation completion. | 2 years
To characterize patient reported outcomes within 1 year of reirradiation using the MDASI BT forms for intracranial tumors. | 1 years
To characterize patient reported outcomes within 1 year of reirradiation using the CTB COMP forms for intracranial tumors. | 1 years
To characterize patient reported outcomes within 1 year of reirradiation using the MDASI SP form for spinal tumors. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The New York Proton Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No